CLINICAL TRIAL: NCT00675181
Title: Effects of Melatonin on Oxygen Consumption and Choroidal Blood Flow in Women With Vasospastic Syndrome in Comparison to Controls
Brief Title: Effects of Melatonin and Oxygen Consumption and Choroidal Blood Flow
Acronym: MelO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 087-KRK-2008-002
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Vasospastic Syndrome
Keywords: melatonin; skin blood flow; choroidal blood flow; vasospastic subjects; normal subjects
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A, 1 (Active Comparator): A, 1 = Melatonin
  Interventions: Drug: Melatonin
- A, 2 (Placebo Comparator): A,2 = Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — 5mg per os
  Arms: A, 1
Drug: Placebo — per os
  Arms: A, 2

SUMMARY:
Does melatonin affect basal metabolic rate, increase choroidal blood flow and reduce the vasospastic syndrome (VS)?

The main questions are:

Do women with VS exhibit...

* a different basal metabolic rate
* a reduced choroidal blood flow
* a reduced increase of oxygen consumption after intake of ice-water
* a different oxygen consumption after melatonin intake
* a different choroidal blood flow after melatonin intake
* a different oxygen consumption after melatonin intake and after intake of ice-water….?

DETAILED DESCRIPTION:
Study description:

Melatonin, a natural hormone of the pineal gland exclusively released during the dark phase, exhibits vasodilatatory effects in distal skin regions and reduces core body temperature. This study investigates whether exogenous melatonin (5mg p.o. at 2p.m.) in the afternoon, when no endogenous melatonin is secreted, increases not only distal skin blood flow, but also choroidal blood flow and changes oxygen consumption. Two subject groups were studied, women with vasospastic syndrome (VS) and controls. The main hypothesis is: melatonin normalizes distal vasoconstriction in VS.

Further questions will also be answered:

Does melatonin affect basal metabolic rate, increase choroidal blood flow and reduce the vasospastic syndrome (VS)?

Do women with VS exhibit:

* a different basal metabolic rate
* a reduced choroidal blood flow
* a reduced increase of oxygen consumption after intake of ice-water
* a different oxygen consumption after melatonin intake
* a different choroidal blood flow after melatonin intake
* a different oxygen consumption after melatonin intake and after intake of ice-water....?

ELIGIBILITY:
Inclusion Criteria:

* vasospastic syndrome
* healthy

Exclusion Criteria:

* sick
* BMI >25 or <18
* migraine
* drug intake

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
-choroidal blood flow -oxygen consumption -Co2 production -skin temperatures -rectal temperatures -blood pressure -eye tension | continously or 2-5 times

CONTACTS AND LOCATIONS:
Overall Officials: Selim Orguel, MD, Study Director — University Eye Clinic, Basel, Switzerland
Locations (1):
- University Eye Clinic, Basel, Switzerland